CLINICAL TRIAL: NCT03600935
Title: Safety and Feasibility of Early Discharge Using the Portico Self-Expanding Prosthesis for Transfemoral Transcatheter Aortic Valve Replacement: The SAFE TAVR Study
Brief Title: Safety and Feasibility of Early Discharge for Transfemoral Transcatheter Aortic Valve Replacement
Acronym: SAFETAVR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: BC Centre for Improved Cardiovascular Health (Other)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBD1
Record Dates: First submitted 2018-07-04; First posted 2018-07-26 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-07

CONDITIONS: Aortic Valve Stenosis
Keywords: Transcatheter Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vancouver Clinical Pathway (Experimental): The Vancouver Clinical Pathway utilizes objective anatomical and functional screening criteria as well as strict peri-procedural guidelines to determine if next day discharge home is appropriate.
  Interventions: Other: Vancouver Clinical Pathway

INTERVENTIONS:
Other: Vancouver Clinical Pathway — Vancouver Clinical Pathway

SUMMARY:
The primary objective of this study is to determine the efficacy, safety and feasibility of next day discharge home in patients undergoing self-expandable transfemoral TAVR utilizing the Vancouver 3M Clinical Pathway.

ELIGIBILITY:
Inclusion Criteria:

Patients with severe symptomatic aortic stenosis undergoing elective transfemoral TAVR with a self-expanding transcatheter heart valve

1. Considered at increased surgical risk by the Multidisciplinary Heart Team
2. Informed written consent

Exclusion Criteria:

1. Non-cardiovascular co-morbidity reducing life expectancy to <3 years
2. Any factor precluding 1 year follow-up
3. Inadequate CT image acquisition to perform area-based annular CT sizing, exclude adverse root features, and determine a coaxial valve deployment angle (CT is not required for valve-in-valve procedures)
4. Predicted inability to perform uncomplicated percutaneous vascular access and closure
5. Illiofemoral diameter <6 mm (for 23 and 25 mm valves) and <6.5 mm (for 27 and 29 mm valves) measured at or below the femoral head
6. Surgical prosthesis <23 mm (labelled size) for valve-in-valve procedure
7. In-patient (unless clinically stable, mobilizing at baseline, and primarily in hospital for logistical reasons)
8. Language barriers (inability to understand peri-procedural and discharge instructions)
9. Insufficient social support post procedure to allow next day discharge
10. Airway unfavourable for emergent intubation
11. Inability to lay supine without conscious sedation or general anaesthetic

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
The composite of all-cause mortality or stroke | 30 days post-procedure
The proportion of patients undergoing elective transfemoral TAVR using the Vancouver Clinical Pathway, who are discharged the next day | Discharge 1 day after procedure

SECONDARY OUTCOMES:
All-cause mortality | 30 days post-procedure
Stroke | 30 days post-procedure
Major vascular complications | 30 days post-procedure
Major/Life-threatening bleed | 30 days post-procedure
Any hospital readmission | 30 days post-procedure
>mild paravalvular regurgiation | Immediately after a procedure is performed or at time immediately prior to discharge, up to 48 hours after procedure
New permanent pacemaker | 30 days post-procedure
Patient is converted from local to general anaesthetic/receives intubation during procedure | This happens during the procedure
Myocardial infarction | This happens during the procedure
Repeat procedure for valve-related dysfunction | 30 days post-procedure
Stage 3 acute kidney injury (need for dialysis) | 30 days post-procedure
Patient-centred outcomes including health related quality of life as measured by KCCQ at baseline, 30 days and 1 year | Baseline, and 30 days and 1 year post-procedure

OTHER OUTCOMES:
Death or stroke | 1 year post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: David A Wood, MD, Principal Investigator — University of British Columbia; John A Webb, MD, Principal Investigator — University of British Columbia